CLINICAL TRIAL: NCT04361604
Title: Clinical Characterisation Protocol for COVID-19 in People Living With HIV
Acronym: COVIDHIV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A00984-35
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Adult Patients Living With HIV (PLWHIV) With Confirmed Infection With SARS-CoV-2 Since 1st January 2020

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Biological collection for the research :
  blood, saliva, rectal swab (stool swab), urine, nasopharyngeal swab, conjonctival swab, semen (for 20 PLWHIV).
  CSF or other samples if indicated as part of standard care requires
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 250 Patients co infected HIV and SRAS-CoV2: Cohort of Patient co infected HIV AND SRAS-CoV2
  Interventions: Biological: Biological collection (patients co infected HIV Sras-CoV-2); Other: Auto-questionnaires (patients co infected HIV Sras-CoV-2); Other: Qualitative interviews (in 40 patients : 20 with COVID-19 and 20 without COVID-19)
- 20 patients infected HIV without COVID-19: Group of 20 comparative patients PLWHIV without COVID-19. This group will realise only the interview of the research.
  Interventions: Other: Qualitative interviews (in 40 patients : 20 with COVID-19 and 20 without COVID-19)

INTERVENTIONS:
Biological: Biological collection (patients co infected HIV Sras-CoV-2) — Biological sampling (blood,saliva, tear urine, stool, respiratory tract, semen only for 20 patients, or other samples if indicated.)
  Groups: 250 Patients co infected HIV and SRAS-CoV2
Other: Auto-questionnaires (patients co infected HIV Sras-CoV-2) — 4 autoquestionnaires will be collected : HADS Hospital anxiety and depression scale, PCL-5 (post-traumatic stress disorder checklist version DSM-5), symptoms with the modified Justice Symptom Index PROQOL-HIV
  Groups: 250 Patients co infected HIV and SRAS-CoV2
Other: Qualitative interviews (in 40 patients : 20 with COVID-19 and 20 without COVID-19) — Qualitative interviews will be realized in 40 patients (20 with COVID-19 and 20 without COVID-19)

SUMMARY:
There is very little data so far to determine whether people living with HIV (PLWHIV) are at greater risk of COVID-19 acquisition or severe disease. HIV infection is associated with deficiencies in both humoral and cell-mediated immunity that could potentially alter the course and severity of common infections. The investigators will study the correlation between clinical and immunovirological data. The singularity of this work is to have an in-depth immunovirological approach linked to the clinical characteristics in COVID-19 HIV co-infected patients. COVIDHIV is the only study to date to offer this combined approach in PLWHIV.

This protocol is a historical and prospective cohort study of PLWHIV presenting COVID-19 The primary objectives are to describe the course of COVID-19 disease in patients infected with HIV

DETAILED DESCRIPTION:
Infectious diseases are a major cause of death worldwide. Recently a new coronavirus named SARS-CoV-2 has been identified as responsible of an initial epidemic respiratory disease, named COVID-19, in China since the 31 December 20191. COVID-19 has developed into a pandemic, with small chains of transmission in many countries and large chains resulting in extensive spread in a some countries, such as Italy, Iran, South Korea, and Japan 2 . Most countries are likely to have spread of COVID-19, at least in the early stages, before any mitigation measures have an impact and the COVID -19 epidemic is gradually taking hold in France 3.

There is very little data so far to determine whether people living with HIV (PLWHIV) are at greater risk of COVID-19 acquisition or severe disease. HIV infection is associated with deficiencies in both humoral and cell-mediated immunity that could potentially alter the course and severity of common infections. Although use of cART partially restores immune system, HIV-infected persons may remain at increased risk for morbidity associated with viral illnesses, especially if the ability to generate antigen-specific responses remains impaired 5. Additional factors, such as the high prevalence of smoking and chronic lung diseases among such patients, may further predispose HIV-infected patients to respiratory tract infections. Finally, they could be considered more vulnerable to SARS-CoV-2 infection because their immune systems are already under strain and cannot avoid the possibility of atypical presentations in these patients. Thus, we would like to implement a research as soon as possible concerning PLWHIV in order to adapt the care of these patients as fast as possible.

The investigator will study the correlation between clinical and immunovirological data. The singularity of this work is to have an in-depth immunovirological approach linked to the clinical characteristics in COVID-19 HIV co-infected patients. COVIDHIV is the only study to date to offer this combined approach in PLWHIV.

This protocol is a historical and prospective cohort study of PLWHIV presenting COVID-19

The primary objectives are to describe the course of COVID-19 disease in patients infected with HIV-1, and more specifically to:

* Describe the clinical and the biological features of the COVID-19 disease in PLWHIV
* Correlate the clinical characteristics with the immunovirological characteristics
* Describe the major complications and determine the factors associated with a worse evolution in PLWHIV
* Compare the data obtained to those of the similar works in progress in non PLWHIV
* Evaluate post-infectious clinical effects at a distance from the acute phase This study will enroll 250 adult patients living with HIV (PLWHIV) with confirmed infection with SARS-CoV-2 since 1st January 2020. Recruitment of patients with Day 1 (enrolment) data is the priority.

Twenty adult patients living with HIV (PLWHIV) without confirmed infection with SARS-CoV-2 will be enrolled only for qualitative interview.

In order to be the most representative of PLHIV population and reach the number of patients to be included people who do not have social security affiliation or who are eligible may be included in the study. A derogation will be requested from the CPP for this.

Research interventions include prospective collection of clinical data and biological sampling (blood, saliva, rectal swab (stool swab), urine, nasopharyngeal swab, conjonctival swab, semen (for 20 PLWHIV), CSF or other samples if indicated as part of standard care.). Auto-Questionnaires will be collected. Qualitative interviews will be realized in 40 patients (20 with COVID-19 and 20 without COVID-19)

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the 250 patients with COVID19

* Patient living with HIV (PLWHIV)
* Patient with confirmed infection with SARS-CoV-2 since 1st January 2020 with and without criteria of hospitalisation.

Inclusion criteria for the 20 patients without COVID19 (who will only realize the qualitative interview)

* Patient living with HIV (PLWHIV)
* Patient who did not have COVID-19

Exclusion Criteria:

Exclusion criteria for the 250 patients with COVID19

* Confirmed diagnosis of another pathogen than SARS-CoV-2
* Refusal by participant, or appropriate representative.
* Being under guardianship or trusteeship mandate for future protection
* Participate to another study without consent of the promoter
* Patients less than 18 years old
* No Beneficiary or entitled to a social security scheme or state medical aid.

Exclusion criteria for the 20 patients without COVID19 (who will only realize the qualitative interview)

* Refusal by participant, or appropriate representative.
* Being under guardianship or trusteeship mandate for future protection
* Participate to another study without consent of the promoter
* Patients less than 18 years old
* No Beneficiary or entitled to a social security scheme or state medical aid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll 250 adult patients living with HIV (PLWHIV) with confirmed infection with SARS-CoV-2 since 1st January 2020. Recruitment of patients with Day 1 (enrolment) data is the priority.
  Twenty adult patients living with HIV (PLWHIV) without confirmed infection with SARS-CoV-2 will be enrolled only for qualitative interview.
  In order to be the most representative of PLHIV population and reach the number of patients to be included people who do not have social security affiliation or who are eligible may be included in the study. A derogation will be requested from the CPP for this.
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Describe the course of COVID-19 disease in patients infected with HIV, | 6 months
  Biological sample collection

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine and Clinical Immunology of Professor Cécile Goujard, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No